CLINICAL TRIAL: NCT04013386
Title: Effects of Aprepitant/Dexamethasone Versus Mertazepine /Dexamethasone on Postoperative Nausea and Vomiting After Laparoscopic Sleeve Surgery: a Randomized Controlled Trial
Brief Title: Effects of Aprepitant/Dexamethasone Versus Mertazepine /Dexamethasone on Postoperative Nausea and Vomiting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dr.Ibrahim Mamdouh Esmat, Assistant Professor of Anesthesia and Intensive Care Department, Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R 36 / 2019
Record Dates: First submitted 2019-07-05; First posted 2019-07-09 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Nausea and Vomiting, Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Aprepitant; Dexamethasone; Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aprepitant/Dexamethasone Group (Active Comparator)
  Interventions: Drug: Aprepitant and Dexamethasone
- Mertazepine /Dexamethasone Group (Active Comparator)
  Interventions: Drug: Mirtazapine and Dexamethasone
- Dexamethasone Group (Active Comparator)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Aprepitant and Dexamethasone — Aprepitant capsule 80 mg and Dexamethasone 8 mg IVI
  Arms: Aprepitant/Dexamethasone Group
Drug: Mirtazapine and Dexamethasone — Mirtazapine tablet 30 mg and Dexamethasone 8 mg IVI
  Arms: Mertazepine /Dexamethasone Group
Drug: Dexamethasone — Dexamethasone 8 mg IVI
  Arms: Dexamethasone Group

SUMMARY:
Laparoscopic sleeve gastrectomy (LSG) is an emerging treatment modality among the various types of surgical approach to obesity (1). The incidence of PONV in obese patients undergoing bariatric surgery, who did not receive antiemetic prophylaxis, is high at nearly 70-80 % (2,3). Postoperatively, bariatric patients appear to suffer from nausea and vomiting more frequently than normal weight or obese patients.

DETAILED DESCRIPTION:
Currently, available interventions for PONV prophylaxis, especially as monotherapy, lack universal efficacy. Use of combination therapies with different pharmacological basis is likely to bring down rates of PONV. (6) Intravenous dexamethasone (8-10mg) reduces the incidence of PONV, minimizing activity of phospholipase A2 and blocking the expression of cyclooxygenase (COX)2 mRNA that reduce production of prostaglandin and control the release of endorphins.

Aprepitant has demonstrated powerful additive effects when combined with dexamethasone and a 5-HT3 to prevent both acute and delayed chemotherapy-induced nausea and vomiting (CINV), and in the prevention of postoperative nausea and vomiting (PONV) The use of mirtazapine in the management of nausea and vomiting has been reported for both treatment and premedication

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II
* Body mass index (BMI) ≥ 35 kg/cm-2

Exclusion Criteria:

* Patients with gastrointestinal disorders,
* Patients with significant major organ disease,
* Patients received antidepressant drugs,
* Patients received an anti-emetic drug within 48 h before surgery,
* Patients on treatment with systemic glucocorticoids within 4 weeks before surgery.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of aprepitant/dexamethasone versus mirtazapine/dexamethasone on PONV prophylaxis after laparoscopic sleeve surgery | First 24 hours(h) postoperative.
  Incidence (%) of nausea and vomiting in 24 hours(h) postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Mohamed Ashoor, MD, Study Director — Faculty of Medicine, Ain- shams University
Locations (1):
- Ain-Shams University Hospitals, Cairo, Egypt

REFERENCES:
- [Derived] Ashoor TM, Kassim DY, Esmat IM. A Randomized Controlled Trial for Prevention of Postoperative Nausea and Vomiting after Laparoscopic Sleeve Gastrectomy: Aprepitant/Dexamethasone vs. Mirtazapine/Dexamethasone. Anesthesiol Res Pract. 2022 Apr 30;2022:3541073. doi: 10.1155/2022/3541073. eCollection 2022. PMID 35535050